CLINICAL TRIAL: NCT04166370
Title: Bangladesh Multisectoral Nutrition Project: Social Protection Mixed Methods Study
Brief Title: Bangladesh MSNP: Social Protection Mixed Methods Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped due to funding
Sponsor: FHI 360 (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1236187; 1432173 (Other: FHI 360)
Record Dates: First submitted 2019-10-15; First posted 2019-11-18 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Stunting; Undernutrition
Keywords: Bangladesh; Multisectoral; Cash Transfer; Randomized
MeSH Terms: conditions — Growth Disorders; Malnutrition

STUDY DESIGN:
Intervention Model Description: cluster-randomized, controlled trial (cRCT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Practice (Active Comparator): Current Standard of Practice
  Interventions: Other: Control
- Strengthened Services and Social Behavioral Change (SBCC) (Experimental): Increase referrals to health services, strengthen health services, and provide enhanced social and behavior change communication (SBCC)
  Interventions: Other: Strengthened (Services and SBCC)
- Strengthened Services and SBCC plus Conditional Cash Transfer (Experimental): Increase referrals to health services, strengthenhealth services, provide enhanced SBCC, as well as cash transfers that are conditional on a mother attending antenatal care (ANC) and monthly nutrition education SBCC group sessions.
  Interventions: Other: Strengthened (Services and SBCC) + CCT

INTERVENTIONS:
Other: Control — The standard of care includes nutrition and health services provided to all pregnant women and mothers of children under-2 as provided by the GoB and their supporting partners. Services that should be provided include clinic-level infant and young child feeding (IYCF) counseling, growth monitoring and promotion, immunization, iron and folic acid distribution for pregnant women, ANC, safe delivery at community and referral for complications, vitamin-A supplements for postpartum women and children, deworming and management of common childhood illness.
  Arms: Standard of Practice
Other: Strengthened (Services and SBCC) — Strengthening referrals to health services- Needed improvements to existing health referral networks will be assessed, identified and implemented. Peer leaders will refer PLW to nearby service delivery points.
  Improving quality of health/nutrition services- Health-related service providers will be trained and supervised on nutrition best practices.
  SBCC- Primarily target PLW. Delivered using traditional and digital channels. Text/voice messages will be sent to PLW twice per week. Family members (e.g. husband) will also be encouraged to sign up for these messages. Female community nutrition promoters will also be deployed; delivering SBCC during group meetings and in health facilities. Mothers' groups will be established, and will be led by peer leaders, mentored in the delivery of messages on nutrition behavior.
  Arms: Strengthened Services and Social Behavioral Change (SBCC)
Other: Strengthened (Services and SBCC) + CCT — Will include all components of the strengthened intervention and participants will receive monthly cash transfers, which is about 25% of monthly consumption expenditure among poor rural households in Bangladesh. Cash transfers will begin when a woman enrolls (at any time during her pregnancy or until 2 months after giving birth). The monthly transfer will continue until a child is 12 months of age, thereby supporting mothers during the critical period of complementary food introduction. The transfer is contingent on having had a minimum of 4 ANC visits and monthly participation in mother's group SBCC sessions.
  Arms: Strengthened Services and SBCC plus Conditional Cash Transfer

SUMMARY:
Despite progress in reducing high levels of undernutrition in Bangladesh, gaps in progress persist. They are particularly acute between rural and urban areas, and between the lowest wealth quintile and highest. According to the 2016 Bangladesh DHS report, 38% of rural children under five were stunted compared to 31% of urban children. Forty-nine percent of children in the lowest wealth quintile were stunted compared to 19% in the highest.

To address these discrepancies and lower the overall level of stunting, research is being conducted to assist the government of Bangladesh (GoB) in determining the most effective ways to reduce levels of stunting. The primary objective of this research is to compare the effectiveness of two multisectoral nutrition intervention packages--one with and without a conditional cash transfer (CCT) component--to the current standard of practice. A cluster-randomized controlled trial using mixed methods will be used to evaluate effectiveness. The two intervention arms are as follows;

* Strengthened: Referrals to health services, strengthened health services, and enhanced social and behavior change communication (SBCC)
* Strengthened + CCT: Referrals to health services, strengthened health services, enhanced SBCC and cash transfers conditional on a mother attending antenatal care (ANC) and monthly nutrition education SBCC group sessions.

The study's primary outcome is the percentage of children 6-23 months old receiving a minimum acceptable diet (MAD), as a proximate determinant for stunting. MAD is defined as the proportion of children 6-23 months old who receive both the minimum feeding frequency and minimum dietary diversity for their age group and breastfeeding status. It will be assessed based on the mother/caregiver report. Secondary outcomes include assessing the knowledge, attitudes, and practices around breastfeeding, complementary feeding, water sanitation and hygiene, health services and gender norms. Quantitative surveys, in depth interviews, focus group discussions, and detailed program monitoring data will be used to assess intervention strengths, weakness, and cost effectiveness.

DETAILED DESCRIPTION:
According to the 2014 Bangladesh Demographic and Health Survey (BDHS), 36% of children under the age of five were stunted, 14% were wasted and 33% were underweight. These results reflect positive trends in stunting and underweight since 2004, though the rate of decline in undernutrition slowed from 2011 to 2014. And, despite positive trends, there remain gaps in key indicators between rural and urban areas and between those in the highest and lowest wealth quintiles. For instance, according to the BDHS, 38% of rural children under five were stunted compared to 31% of urban children. The wealth discrepancies are even greater; 49% of children under five in the lowest wealth quintile were stunted compared to 19% in the highest quintile.

In 2017, the GoB approved the second National Plan of Action for Nutrition (NPAN 2) 2016-2025. The plan aims to improve nutrition and eliminate malnutrition, with a focus on children, adolescent girls, and pregnant and lactating women. Specific targets of NPAN 2 include reducing stunting to 25% among children under 5; reducing wasting to less than 8% and reducing underweight to less than 15%. A significant acceleration in the annual rate of reduction to 3.3% needs to occur in order to achieve the ambitious Targets by 2025. This acceleration requires high-level political commitment, a strong policy framework, effective coordinating mechanisms, adequate resourcing, strong involvement of local civil society groups, and high impact, cost-effective, multisectoral nutrition interventions.

In 2017, USAID awarded FHI 360 the Strengthening Multisectoral Nutrition Programming through Implementation Science Activity (hereafter referred to as "the Project") to test and refine multisectoral nutrition approaches in high stunting areas of Bangladesh. Under the Project, research is being conducted to assess the effect of different multisectoral nutrition intervention packages aimed at improving nutrition outcomes that are known to contribute to overall healthy nutritional status of children under two in Bangladesh. One of the intervention packages studied by the Project focuses on conditional cash transfers (CCT) for social protection. The primary objective of this study is to compare the effectiveness of the current standard of practice with two multisectoral intervention packages--one with and without a CCT intervention. The two intervention arms are as follows:

* Strengthened: Referrals to health services, strengthened health services, and enhanced social and behavior change communication (SBCC)
* Strengthened + CCT: Referrals to health services, strengthened health services, enhanced SBCC and cash transfers conditional on a mother attending antenatal care (ANC) and monthly nutrition education SBCC group sessions.

A cluster-randomized, controlled trial (cRCT) design will be used to evaluate effectiveness. The interventions will be delivered at the level of the union, which is a geo-political unit with an average population of 25,000 people. A total of 60 unions in Khulna and Barishal Divisions of Bangladesh will be randomly allocated to one of the three study arms: Control (Current Practice), Strengthened Intervention, or Strengthened + CCT Intervention. Outcome data will be collected through face-to-face interviews using structured questionnaires with independently selected random samples of mothers/caregivers of children ages 6 to 23 months at baseline (pre-intervention) and again at endline. At both timepoints, participants will be chosen from a sub-sample of the general population who meet the eligibility criteria. Baseline data will be conducted prior to initiation of study activities. Endline data collection will be conducted after two years.

A process evaluation will be completed between baseline and endline to understand how well the interventions were implemented, their costs, and ways they may be improved.

The final evaluation analysis of the cRCT to be done at endline, and will focus on comparing the effect of the intervention on the study outcomes. The study's primary outcome is the percentage of children 6-23 months old receiving a minimum acceptable diet (MAD), as a proximate determinant for stunting. MAD is defined as the proportion of children 6-23 months old who receive both the minimum feeding frequency and minimum dietary diversity for their age group and breastfeeding status. It will be assessed based on the mother/caregiver report. Secondary outcomes include assessing the knowledge, attitudes, and practices around breastfeeding, complementary feeding, water sanitation and hygiene, health services and gender norms.

It is anticipated an analysis of covariance (ANCOVA) approach will be used for a post-only comparison of study arms with possible adjustment for baseline levels in an aggregate manner (note: aggregation for baseline adjustment will be needed given the independent samples selected at each time point). Generalized mixed models to compare the study groups and adjust for clustering at the union level will be used. A logit link will be used for the primary outcome (i.e., minimum acceptable diet) as it is a dichotomous outcome, while other link functions will be used for other outcomes as appropriate. It is hypothesized that the intervention arm with the enhanced SBCC will be superior to standard practice. It is further hypothesized that adding CCT along with the enhanced SBCC will produce an even greater effect. These pairwise comparisons will be tested using the model parameter estimates.

ELIGIBILITY:
Inclusion Criteria:

* mother/caregiver of child 6-23 months of age
* Child 6-23 months is mothers 1st or second (living) child
* resides in an extreme poor household, which is defined in Barishal as less than BDT 1778/month on household expenditures or in Khulna as less than BDT 1677/month on household expenditures

Note: study inclusion criteria is different from intervention enrollee criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-26 (Actual); Primary Completion 2020-06-28 (Actual); Study Completion 2020-06-28 (Actual)

PRIMARY OUTCOMES:
Change in the proportion of Children 6-23 months receiving Minimum Acceptable Diet based on mother/caregiver report | This outcome will be assessed not earlier than 22 months after the introduction of the interventions
  Minimum Acceptable Diet (MAD) is defined as children by WHO as the proportion of children 6-23 months of age who receive both the minimum feeding frequency and minimum dietary diversity for their age group and breastfeeding status

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Hoke, PhD, Principal Investigator — FHI 360; Taufique Jorder, DrPH, Principal Investigator — FHI 360
Locations (1):
- FHI 360, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared in accordance with USAID's open data policy.
Time Frame: Approximately January 2022.
Access Criteria: Data will be made available upon request, submitted with a brief concept describing intended use of data.

REFERENCES:
- [Background] BNNC (2017). Second National Plan of Action on Nutrition. Dhaka. Bangladesh National Nutrition Council (BNNC), 2017.
- [Background] Ahmed AU, et al. Which Kinds of Social Safety Net Transfers Work Bets for the Ultra Poor in Bangladesh? Operation and Impacts of the Transfer Modality Research Initiative. Dhaka, IFPRI and WFP, 2016.
- [Background] BBS (2017). Preliminary Report on Household Income and Expenditure Survey 2016. Dhaka, Bangladesh Bureau of Statistics (BBS), 2017.
- [Background] Black RE, Victora CG, Walker SP, Bhutta ZA, Christian P, de Onis M, Ezzati M, Grantham-McGregor S, Katz J, Martorell R, Uauy R; Maternal and Child Nutrition Study Group. Maternal and child undernutrition and overweight in low-income and middle-income countries. Lancet. 2013 Aug 3;382(9890):427-451. doi: 10.1016/S0140-6736(13)60937-X. Epub 2013 Jun 6. PMID 23746772
- [Background] Black RE, Allen LH, Bhutta ZA, Caulfield LE, de Onis M, Ezzati M, Mathers C, Rivera J; Maternal and Child Undernutrition Study Group. Maternal and child undernutrition: global and regional exposures and health consequences. Lancet. 2008 Jan 19;371(9608):243-60. doi: 10.1016/S0140-6736(07)61690-0. No abstract available. PMID 18207566
- [Background] FHI 360 (2016). SHIKHA Project Final Report. Dhaka, Bangladesh: FHI 360.
- [Background] Food and Nutrition Technical Assistance III Project (FANTA). 2017. Multisectoral Nutrition Programming: FANTA Achievements and Lessons Learned. Washington, DC: FHI 360/ FANTA.
- [Background] GoB. Bangladesh 2nd National Plan of Action (NPAN2) 2016-2025. 2015. Dhaka, Government of Bangladesh.
- [Background] Islam F. National Social Security Strategy (NSSS): Progress of Action Plan preparation. Presented at the Technical Symposium on Nutrition Sensitive Social Protection in Bangladesh, December 2017.
- [Background] MI. (2009). Investing in the future: A united call to action on vitamin and mineral deficiencies: Micronutrient Initiative
- [Background] National Institute of Population Research and Training (NIPORT), Mitra and Associates, and ICF International. 2016. Bangladesh Demographic and Health Survey 2014. Dhaka, Bangladesh, and Rockville, Maryland, USA: NIPORT, Mitra and Associates, and ICF International
- [Background] Save the Children (2012). Nutrition in the First 1000 Days: State of the World's Mothers 2012 Save the Children
- [Background] WHO (2008). Indicators for assessing infant and young child feeding practices, part 1: definitions
- [Background] Essential Nutrition Actions: Improving Maternal, Newborn, Infant and Young Child Health and Nutrition. Geneva: World Health Organization; 2013. Available from http://www.ncbi.nlm.nih.gov/books/NBK258736/ PMID 25473713
- [Background] WHO, UNICEF, and USAID. (2015). Improving Nutrition Outcomes with Better Water, Sanitation and Hygiene: Practical Solutions for Policies and Programmes. Switzerland: WHO
- See also: UNICEF. (2018). Child malnutrition estimates — http://data.unicef.org/topic/nutrition/malnutrition